CLINICAL TRIAL: NCT03763175
Title: Evaluation of the Efficacy and Safety of Single, Daily Oral Doses of SYN-010 Compared to Placebo in Adult Patients With Irritable Bowel Syndrome With Constipation (EASE-DO)
Brief Title: Efficacy and Safety of SYN-010 in IBS-C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim Futility Analysis
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Theriva Biologics, Inc. (Industry)
Responsible Party: Principal Investigator, Ali Rezaie, MD, Director of GI Motility, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 54792
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Irritable Bowel Syndrome with Constipation; Lovastatin; SYN-010
MeSH Terms: interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SYN-010 21 mg (Active Comparator): Enrolled subjects will be screened and randomized into the three study arms in a 1:1:1 ratio. 50 subjects with constipation-predominant irritable bowel syndrome (IBS-C) will be administered a 12-week course of lovastatin (21 mg PO QD). Study activities will be the same across all three arms.
  Interventions: Drug: SYN-010 21 mg
- SYN-010 42 mg (Active Comparator): Enrolled subjects will be screened and randomized into the three study arms in a 1:1:1 ratio. 50 subjects with constipation-predominant irritable bowel syndrome (IBS-C) will be administered a 12-week course of lovastatin (42 mg PO QD). Study activities will be the same across all three arms.
  Interventions: Drug: SYN-010 42 mg
- Placebo (Placebo Comparator): Enrolled subjects will be screened and randomized into the three study arms in a 1:1:1 ratio. 50 subjects with constipation-predominant irritable bowel syndrome (IBS-C) will be administered a 12-week course of placebo. Study activities will be the same across all three arms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYN-010 21 mg — 21 mg lovastatin will be administered to patients diagnosed with IBS-C to evaluate whether the medication and dose is effective in increasing frequency of completely spontaneous bowel movements. The secondary objectives of the study are to assess the role of lovastatin lactone in increasing overall stool frequency and reducing abdominal pain severity, bloating severity, and rescue medication use. Additional endpoints include improvement in reported adequate relief and the effect of the study drug in lowering exhaled methane levels.
  Other Names: lovastatin
  Arms: SYN-010 21 mg
Drug: SYN-010 42 mg — 42 mg lovastatin will be administered to patients diagnosed with IBS-C to evaluate whether the medication and dose is effective in increasing frequency of completely spontaneous bowel movements. The secondary objectives of the study are to assess the role of lovastatin lactone in increasing overall stool frequency and reducing abdominal pain severity, bloating severity, and rescue medication use. Additional endpoints include improvement in reported adequate relief and the effect of the study drug in lowering exhaled methane levels.
  Other Names: lovastatin
  Arms: SYN-010 42 mg
Drug: Placebo — A placebo will be administered to patients diagnosed with IBS-C to evaluate whether the medication and dose is effective in increasing frequency of completely spontaneous bowel movements. The secondary objectives of the study are to assess the role of lovastatin lactone in increasing overall stool frequency and reducing abdominal pain severity, bloating severity, and rescue medication use. Additional endpoints include improvement in reported adequate relief and the effect of the study drug in lowering exhaled methane levels.
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is a gastrointestinal (GI) syndrome characterized by chronic abdominal pain and altered bowel habits in the absence of any organic cause. The symptoms of IBS not only adversely affect a patient's health-related quality of life (QoL), but also place a significant financial burden on society due to reduced work productivity and increased use of healthcare-related resources. Patients with IBS frequently complain of abdominal bloating and increased gas production in the form of flatulence or belching. The prevalence in North America and Europe is approximately 10-15%. Irritable bowel syndrome affects all ages and genders however there is a 2:1 female predominance in North America. Irritable bowel syndrome is classified into 4 subtypes based on stool pattern: IBS with constipation (IBS-C), IBS with diarrhea, mixed IBS, and un-subtyped IBS. Irritable bowel syndrome with constipation is defined as the presence of hard or lumpy stools with ≥ 25 percent of bowel movements and loose or watery stools with < 25% of bowel movements.

SYN-010 is a modified release, oral formulation of lovastatin being developed for the treatment of IBS-C. The SYN-010 program is based predominantly on research by Dr. Mark Pimentel and collaborators hypothesizing that reduction in intestinal methane (methane) production can reverse constipation and improve global symptoms in IBS-C. Methane production in humans is due to methanogenic archaea in the intestine, predominantly Methanobrevibacter smithii (M. smithii). Methane, the key product of anaerobic respiration of methanogens, had been perceived to produce no ill effects in humans aside from gaseous distention. However, several research groups worldwide have shown that a significant percentage of patients with IBS-C excrete methane, and elevated methane production by methanogens correlates with constipation and related symptoms in both IBS-C and chronic idiopathic constipation. A direct causative role for methane in IBS-C was demonstrated in a recent case report, wherein a woman undergoing fecal microbiota transplantation (FMT) for C. difficile infection unknowingly received stool containing a high concentration of methanogens. The FMT recipient rapidly developed severe symptoms of IBS-C that were subsequently reversed by ablation of methane production.

DETAILED DESCRIPTION:
SYN-010 has previously been evaluated in consecutive Phase 2a clinical trials. Sixty-three (63) IBS-C patients with high breath methane (>10 ppm) at screening were enrolled in a multicenter, randomized, controlled, double-blinded clinical trial (RCT) in which they received SYN-010 21 mg, SYN-010 42 mg or Placebo once daily for 4 weeks. Fifty-four (54) subjects who completed the RCT continued into an open-label extension (EXT) in which all subjects received SYN-010 42 mg once daily for an additional 8 weeks.

The SYN-010 Phase 2a studies were intentionally designed as mechanistic proof-of-concept studies, wherein reductions in breath methane were employed as a rapid and cost-effective means by which to determine if SYN-010 could be effective in treating an underlying cause of symptoms in IBS-C. Breath methane was reduced relative to baseline in SYN-010 treatment groups, and lower breath methane levels correlated with an increased number of complete spontaneous bowel movements (CSBMs) at week 12, consistent with the proposed methane-inhibiting action of lovastatin lactone.

Since lovastatin has not previously been used to treat IBS-C patients, the SYN-010 Phase 2a studies were also focused on the safety of the SYN-010 dosage form. Daily doses of SYN-010 were well-tolerated by IBS-C patients over the 12-week treatment period (at least 8 weeks of SYN-010 42 mg). SYN-010 did not cause clinically meaningful or persistent changes in serum liver and muscle markers in IBS-C patients at daily doses of 21 mg and 42 mg. Modest decreases from baseline in lipid parameters observed after 7 days of SYN-010 21 mg or 42 mg had largely faded by 28 days and were not evident after 12 weeks of dosing. Very few adverse events were reported over 12 weeks of SYN-010 treatment and all were of mild or moderate intensity. No serious adverse events were reported and there were no incidences of drug-related diarrhea, which is an important potential benefit of SYN-010 as an IBS-C therapy.

Although the Phase 2a studies were not prospectively powered for formal statistical evaluation of clinical endpoints, compelling improvements in CSBMs, abdominal pain, and bloating were observed in SYN-010 treatment groups. These clinical findings have been presented in multiple public forums and a panel of clinical advisors affirmed that the Phase 2a data validate the need to evaluate optimal dosing of SYN-010 in a larger patient population over a longer dosing period.

Based on the potential clinical benefit observed in Phase 2a, this Phase 2b clinical study will evaluate in more detail the clinical effects of two dose strengths of SYN-010 administered over a longer treatment period (12 weeks per FDA guidelines) to a larger number of IBS-C patients. The study will seek more definitive evidence regarding potential symptom improvements and safety in IBS-C patients. The study also seeks to provide new information of relevance to both efficacy and safety by measuring changes to the microbiome in patient stool samples; serum level of cytokine markers of inflammation; and expanded breath gas measurements.

SYN-010 is a hydroxypropyl methylcellulose (HPMC) capsule filled with enteric-coated tablets from which lovastatin is released at different intestinal pH values. The tablets are designed to pass through the stomach unchanged then release a small amount of lovastatin into the duodenum and the majority of the lovastatin dose into the ileocecal junction and colon. The amount of lovastatin to be released into the small and large intestine is anticipated to be consistent with the relative levels of methane-producing archaea in each location of the intestine.

Methane production (methanogenesis) is a ubiquitous process in the human intestine, disposing of hydrogen and other by-products formed during bacterial fermentation. Methane production in humans is almost entirely due to the archeon M. smithii. Elevated intestinal methane production reduces intestinal motility and is a cause of constipation, pain and bloating in IBS-C.

Interest in lovastatin as a potential inhibitor of methanogenesis originated with recognition that the rate-limiting step in the synthesis of archaeal lipid membranes is catalyzed by HMG-CoA reductase (HMGR) which is the target enzyme for cholesterol-lowering statins. Subsequent in vitro studies (described above) and computational studies have since determined that HMGR is not the target for lovastatin anti-methanogenic activity; rather, lovastatin lactone appears to exert a direct effect on methanogenesis enzymes. The mechanism by which lovastatin lactone inhibits methane production by M. smithii has not been conclusively determined; however, detailed computational studies showed that lovastatin lactone may competitively inhibit F420-dependent methylenetetrahydromethanopterin dehydrogenase (mtd), an enzyme that is integral to the M. smithii methanogenesis pathway.

Methanogenic archaea reside predominantly in the human colon, with lower methanogen levels measured in the small intestine of some patients. Methane production at both sites contributes to reduced gastrointestinal motility and rat studies suggest that the ileocecal region may be of particular significance. SYN-010 utilizes a dual-pulse release profile to deliver a portion of the lovastatin dose to the small intestine and the majority of the dose to the ileocecal junction and colon where the most methane-producing organisms are found; the relative amounts of lovastatin released into the small and large intestine are consistent with the anticipated relative levels of methanogens in each location.

Lovastatin lactone exerts its methane-reducing effect in the intestinal lumen and systemic absorption of lovastatin is not required for its therapeutic effect in IBS-C.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged between 18 and 65 years inclusive.
* Patient must be willing and able to participate in the study for the required duration, understand and sign the informed consent (ICF), and be willing to comply with all protocol-related visits and procedures.
* Patient has had IBS-C symptoms (as defined by Rome III diagnostic criteria) for at least 6 months prior to diagnosis.
* Patient has an average score of ≥ 3.0 for daily abdominal pain at its worst (11-point numerical rating scale [NRS]) during and up to the 17 days immediately before randomization (i.e. Pre-treatment Period).
* Patient has an average of ≤ 3 CSBMs per week or ≤ 5 SBMs per week during the 17 days immediately before randomization (i.e. Pre-treatment Period).
* Patient has a breath methane level ≥ 10 ppm on a lactulose breath test administered at Screening.
* Patient may be on a stable, continuous regimen of fiber or probiotics one month before the Screening Visit; however, they must maintain a stable dose regimen through Week 12.
* Patient must agree to refrain from starting a new diet, changing stable dose of supplemental fiber, or changing exercise pattern that may affect IBS-C symptoms from the time of Screening through the end of the study. If the patient takes food products that are strong inhibitors of cytochrome P450 3A (CYP3A) (e.g. grapefruit juice, Seville orange juice, St. John's Wort), he/she must agree to refrain from taking these from the time of Screening through the end of the study.
* Patient must agree to use an acceptable method of contraception from the time of signing the ICF to 30 days after the final dose of study drug if the patient is a sexually active female of child-bearing potential (defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause). Adequate contraceptive measures include: oral contraceptives (stable use for two or more cycles before Screening); intrauterine device; Depo-Provera®; Norplant® System implants; partner with a vasectomy; double-barrier birth control (e.g. use of a condom plus diaphragm or condom plus either contraceptive sponge, foam, or jelly); or abstinence. According to drug research standards, male patient must agree to use an acceptable method of contraception and refrain from donating sperm from the time of signing the ICF to 90 days after the final dose of study drug.
* A female patient of child-bearing potential must be non-pregnant and non-lactating and have negative pregnancy tests at the Screening Visit and on Day 1 prior to dosing with study drug.
* Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Willing and able to comply with the protocol, including follow-up visits and examinations.

Exclusion Criteria:

* Patient has loose (mushy) or watery stools for > 25% of their bowel movements (BMs) during the 12 weeks before Screening or during the Screening and Pre-treatment Periods.
* Patient has a history of cathartic colon, laxative, or enema abuse.
* Patient has a history of ischemic colitis.
* Patient has a history of pelvic floor dysfunction.
* Patient has a history of bariatric surgery for the treatment of obesity.
* Patient has a history of surgery to remove a segment of the gastrointestinal (GI) tract at any time before the Screening Visit.
* Patient has any history of myopathy, rhabdomyolysis, chronic myalgia, or familial history of hereditary muscular disorders.
* Patient has been diagnosed with or has a family history of familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer, or any other form of familial colorectal cancer.
* Patient currently has any structural abnormality of the GI tract or a disease or condition that can affect GI motility, or any unexplained and clinically significant symptoms such as lower GI bleeding, rectal bleeding, heme-positive stool, iron-deficiency anemia, weight loss, or systemic signs of infection.
* Patient has had any previous surgery involving the abdomen, pelvis, or retroperitoneal region during the last 12 months prior to Screening, with the exclusion of laparoscopic gallbladder surgery or appendix removal.
* Patient has a history of diverticulitis or any chronic condition that could be associated with abdominal pain or discomfort and could confound the assessments in the study (e.g. inflammatory bowel disease, chronic pancreatitis, polycystic kidney disease, ovarian cysts, endometriosis, or lactose intolerance).
* Patient has history of severe renal insufficiency defined as an actual or estimated glomerular filtration rate of < 30 mL/min/1.73 m2 within the 6 months prior to Screening Visit.
* Patient has any history of a medical condition or a concomitant medical condition that, in the opinion of the investigator, would compromise the patient's ability to complete the study safely or could confound the assessments in this study (e.g. uncontrolled hypothyroidism).
* Patient is known to have elevated liver enzyme levels (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP]) or creatine kinase levels that are ≥ 1.5 times the upper limit of normal (ULN) that have not been resolved within the 4 weeks prior to consent and/or these elevated levels are present at the Screening Visit laboratory assessment.
* Patient has any abnormal laboratory results, electrocardiogram (ECG) findings, or physical examination findings deemed clinically significant by the investigator during the Screening Period.
* Within 14 days prior to the Screening Visit, patient has used concomitant medications that are: (1) moderate-to-strong inhibitors of cytochrome P450 3A (CYP3A) and/or organ anion transporting polypeptide (OATP)1B1 (e.g. cyclosporine, verapamil, dronedarone, diltiazem, amiodarone, itraconazole, ketoconazole, posaconazole, voriconazole, clarithromycin, telithromycin, human immunodeficiency virus protease inhibitors, boceprevir, telaprevir, nefazodone, erythromycin, cobicistat-containing products); (2) other concomitant medications that are excluded from the lovastatin label (e.g. rifampin, colchicine, ranolazine); or (3) metformin or GLP-1 agonists. Patients should not take any of these concomitant medications during the treatment phase of the study without contacting the investigator.
* Patient has hypersensitivity to statins; or has used any statins, fibrates, > 1 g/day of niacin, or gemfibrozil within the 3 months prior to the Screening Visit.
* Patient reports current chronic or frequent use of drugs known to cause constipation (e.g. narcotics) for the 3 months prior to Screening.
* Patient has taken over-the-counter IBS treatments (e.g. laxatives) or proton pump inhibitors within 3 days prior to the Screening Visit.
* Certain drugs used for the treatment of IBS (e.g. low dose tricyclic antidepressants) may be allowed at the discretion of the Medical Monitor provided the patient remains on a stable dose for one month prior to the Screening Visit and throughout the study with the exception of tegaserod, lubiprostone, linaclotide, metoclopramide, prucalopride, domperidone, or antibiotics within 2 months prior to the Screening Visit. Certain drugs used for the treatment of IBS (e.g. low dose tricyclic antidepressants) may be allowed at the discretion of the Medical Monitor provided the patient remains on a stable dose for one month prior to the Screening Visit and throughout the study with the exception of tegaserod, lubiprostone, linaclotide, metoclopramide, prucalopride, domperidone, CandiBactin, Atrantil, Allimax/Allimed within 2 weeks prior to the Screening Visit or antibiotics within 2 months prior to the Screening Visit.
* Patient has used an opioid chronically or frequently within the 3 months prior to the Screening Visit and for the duration of the study.
* Patient is currently enrolled in, or plans to enroll in, another clinical study or has used any investigational drug or device within 1 month before signing the ICF through the completion of the study.
* Patient has previously participated in a SYN-010 study.
* Patient has a history of alcohol or drug abuse within the 12 months prior to the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezaie, MD MSc, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Cash B, Sullivan S, Barghout V. Total costs of IBS: employer and managed care perspective. Am J Manag Care. 2005 Apr;11(1 Suppl):S7-16. PMID 15926759
- [Background] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866
- [Background] Hungin AP, Whorwell PJ, Tack J, Mearin F. The prevalence, patterns and impact of irritable bowel syndrome: an international survey of 40,000 subjects. Aliment Pharmacol Ther. 2003 Mar 1;17(5):643-50. doi: 10.1046/j.1365-2036.2003.01456.x. PMID 12641512
- [Background] Drossman DA, Dumitrascu DL. Rome III: New standard for functional gastrointestinal disorders. J Gastrointestin Liver Dis. 2006 Sep;15(3):237-41. PMID 17013448
- [Background] American College of Gastroenterology Task Force on Irritable Bowel Syndrome; Brandt LJ, Chey WD, Foxx-Orenstein AE, Schiller LR, Schoenfeld PS, Spiegel BM, Talley NJ, Quigley EM. An evidence-based position statement on the management of irritable bowel syndrome. Am J Gastroenterol. 2009 Jan;104 Suppl 1:S1-35. doi: 10.1038/ajg.2008.122. No abstract available. PMID 19521341
- [Background] Talley NJ, Zinsmeister AR, Van Dyke C, Melton LJ 3rd. Epidemiology of colonic symptoms and the irritable bowel syndrome. Gastroenterology. 1991 Oct;101(4):927-34. doi: 10.1016/0016-5085(91)90717-y. PMID 1889716
- [Background] Pimentel M, Gunsalus RP, Rao SSC, Zhang H. Methanogens in human health and disease. Am J Gastroenterol. 2012 Jul;1(1) Suppl:28-33.
- [Background] Pimentel M, Mayer AG, Park S, Chow EJ, Hasan A, Kong Y. Methane production during lactulose breath test is associated with gastrointestinal disease presentation. Dig Dis Sci. 2003 Jan;48(1):86-92. doi: 10.1023/a:1021738515885. PMID 12645795
- [Background] Kunkel D, Basseri RJ, Makhani MD, Chong K, Chang C, Pimentel M. Methane on breath testing is associated with constipation: a systematic review and meta-analysis. Dig Dis Sci. 2011 Jun;56(6):1612-8. doi: 10.1007/s10620-011-1590-5. Epub 2011 Feb 1. PMID 21286935
- [Background] Furnari M, Savarino E, Bruzzone L, Moscatelli A, Gemignani L, Giannini EG, Zentilin P, Dulbecco P, Savarino V. Reassessment of the role of methane production between irritable bowel syndrome and functional constipation. J Gastrointestin Liver Dis. 2012 Jun;21(2):157-63. PMID 22720304
- [Background] Ghoshal U, Shukla R, Srivastava D, Ghoshal UC. Irritable Bowel Syndrome, Particularly the Constipation-Predominant Form, Involves an Increase in Methanobrevibacter smithii, Which Is Associated with Higher Methane Production. Gut Liver. 2016 Nov 15;10(6):932-938. doi: 10.5009/gnl15588. PMID 27458176
- [Background] Lee KM, Paik CN, Chung WC, Yang JM, Choi MG. Breath methane positivity is more common and higher in patients with objectively proven delayed transit constipation. Eur J Gastroenterol Hepatol. 2013 Jun;25(6):726-32. doi: 10.1097/MEG.0b013e32835eb916. PMID 23395994
- [Background] Suri J, Kataria R, Malik Z, Parkman HP, Schey R. Elevated methane levels in small intestinal bacterial overgrowth suggests delayed small bowel and colonic transit. Medicine (Baltimore). 2018 May;97(21):e10554. doi: 10.1097/MD.0000000000010554. PMID 29794732
- [Background] Chang BW, Rezaie A. Irritable Bowel Syndrome-Like Symptoms Following Fecal Microbiota Transplantation: A Possible Donor-Dependent Complication. Am J Gastroenterol. 2017 Jan;112(1):186-187. doi: 10.1038/ajg.2016.472. No abstract available. PMID 28050036
- [Background] Park YM, Lee YJ, Hussain Z, Lee YH, Park H. The effects and mechanism of action of methane on ileal motor function. Neurogastroenterol Motil. 2017 Sep;29(9). doi: 10.1111/nmo.13077. Epub 2017 Apr 18. PMID 28417537
- [Background] Pimentel M, Lin HC, Enayati P, van den Burg B, Lee HR, Chen JH, Park S, Kong Y, Conklin J. Methane, a gas produced by enteric bacteria, slows intestinal transit and augments small intestinal contractile activity. Am J Physiol Gastrointest Liver Physiol. 2006 Jun;290(6):G1089-95. doi: 10.1152/ajpgi.00574.2004. Epub 2005 Nov 17. PMID 16293652
- [Background] Jahng J, Jung IS, Choi EJ, Conklin JL, Park H. The effects of methane and hydrogen gases produced by enteric bacteria on ileal motility and colonic transit time. Neurogastroenterol Motil. 2012 Feb;24(2):185-90, e92. doi: 10.1111/j.1365-2982.2011.01819.x. Epub 2011 Nov 20. PMID 22097886
- [Background] Mevacor® (lovastatin) tablets. Prescribing information, 2014. Merck & Co., Inc., Whitehouse Station, NJ 08889, USA.
- [Background] Duggan DE, Chen IW, Bayne WF, Halpin RA, Duncan CA, Schwartz MS, Stubbs RJ, Vickers S. The physiological disposition of lovastatin. Drug Metab Dispos. 1989 Mar-Apr;17(2):166-73. PMID 2565206
- [Background] Marsh E, Morales W, Chua KS, Marsh Z, Weitsman S, Wacher V, Kim JH, Pimentel, M. (2015) [Abstract 1771] Lovastatin lactone inhibits methane production in human stool homogenates. Am J Gastroenterol. 110 (Suppl. 1): S753.
- [Background] Morales W, Marsh E, Yu A, Marsh Z, Weitsman S, Barlow GM, Rezaie A, Chang C, Wacher V, Pimentel, M. (2015) [Abstract Mo 2051] Lovastatin improves stool form in Methanobrevibacter smithii colonized rats with constipation. Gastroenterology 148 (Suppl. 1): S-779-80
- [Background] Gottlieb K, Wacher V, Sliman J, Coughlin O, McFall H, Rezaie A, Pimentel M. (2016) [Abstract Su1210] SYN-010, a proprietary modified-release formulation of lovastatin lactone, lowered breath methane and improved stool frequency in patients with IBS-C: results of a multi-center randomized double-blind, placebo-controlled Phase 2a trial. Gastroenterology 150 (Suppl. 1): S496-7.
- [Background] Wacher V, Gottlieb K, Sliman J, Coughlin O, Kokai-Kun, J, McFall H, Pimentel M (2016) [Abstract 562] SYN-010 modified-release lovastatin does not significantly alter lipid parameters at doses that reduce methane and alleviate symptoms in patients suffering irritable bowel syndrome with constipation (IBS-C). Am J Gastroenterol. 111 (Suppl. 1): S256.
- [Background] Hubert S, Chadwick A, Wacher V, Coughlin O, Kokai-Kun J, Bristol A. Development of a Modified-Release Formulation of Lovastatin Targeted to Intestinal Methanogens Implicated in Irritable Bowel Syndrome With Constipation. J Pharm Sci. 2018 Feb;107(2):662-671. doi: 10.1016/j.xphs.2017.09.028. Epub 2017 Oct 6. PMID 28989013
- [Background] Muskal SM, Sliman J, Kokai-Kun J, Pimentel M, Wacher V, Gottlieb K. Lovastatin lactone may improve irritable bowel syndrome with constipation (IBS-C) by inhibiting enzymes in the archaeal methanogenesis pathway. F1000Res. 2016 Apr 8;5:606. doi: 10.12688/f1000research.8406.3. eCollection 2016. PMID 27347377
- [Background] Camilleri M, Lembo AJ, Lavins BJ, MacDougall JE, Carson RT, Williams VS, Nelson LM, Shiff SJ, Currie MG, Kurtz CB, Johnston JM. Comparison of adequate relief with symptom, global, and responder endpoints in linaclotide phase 3 trials in IBS-C. United European Gastroenterol J. 2015 Feb;3(1):53-62. doi: 10.1177/2050640614555946. PMID 25653859
- [Background] Passos MC, Lembo AJ, Conboy LA, Kaptchuk TJ, Kelly JM, Quilty MT, Kerr CE, Jacobson EE, Hu R, Friedlander E, Drossman DA. Adequate relief in a treatment trial with IBS patients: a prospective assessment. Am J Gastroenterol. 2009 Apr;104(4):912-9. doi: 10.1038/ajg.2009.13. Epub 2009 Mar 17. PMID 19293784
- [Derived] Villanueva-Millan MJ, Leite G, Wang J, Morales W, Parodi G, Pimentel ML, Barlow GM, Mathur R, Rezaie A, Sanchez M, Ayyad S, Cohrs D, Chang C, Rashid M, Hosseini A, Fiorentino A, Weitsman S, Chuang B, Chang B, Pichetshote N, Pimentel M. Methanogens and Hydrogen Sulfide Producing Bacteria Guide Distinct Gut Microbe Profiles and Irritable Bowel Syndrome Subtypes. Am J Gastroenterol. 2022 Dec 1;117(12):2055-2066. doi: 10.14309/ajg.0000000000001997. Epub 2022 Sep 6. PMID 36114762

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Started | 20 | 19 | 20
Completed | 19 | 17 | 19
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 20 | 59
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 15 | 45
  Male | 4 | 5 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 19 | 17 | 18 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 19 | 17 | 15 | 51
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average Number of Completely Spontaneous Bowel Movements (CSBM) Compared to the 12-week Treatment Period
Description: Subjects will record their daily bowel movements throughout the duration of the study. Change in weekly average number of CSBMs will be evaluated by comparing reported values pre- and post-treatment.
Time Frame: After completing 12-week course of SYN-010
Population: Change from baseline in weekly average number of CSBMs at Weeks 1 through 12. Weekly average number of CSBMs = 7 x (sum of daily number of CSBMs)/ (number of days with CSBM assessment) for the specific week.
  The analysis for the primary endpoint was performed using the analysis of covariance (ANCOVA) with treatment group and the baseline value as covariates based on the full analysis set. The primary analysis was conducted using the observed values.
Measure: Least Squares Mean (Standard Error); unit: Weekly average CSBMs
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 20
Weekly average CSBMs | 1.53 (0.32) | 0.32 (0.32) | 0.51 (0.33)

2. Secondary Outcome: Proportion of Overall Responders During the 12-week Treatment Period
Description: An overall 12-week responder is defined as a patient with a weekly response in at least 50% of the weeks of treatment (6 of 12 weeks). A weekly response is defined as a decrease in the patient's weekly average score for worst abdominal pain in the past 24 hours of at least 30% compared to baseline and a stool frequency increase of 1 or more CSBMs per week compared with baseline.
Time Frame: After completing 12-week course of SYN-010
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 20
Participants | 1 | 2 | 6

3. Secondary Outcome: Proportion of Overall Stool Frequency Responders During the 12-week Treatment Period
Description: An overall stool frequency responder is defined as a patient with a weekly stool frequency response in at least 50% of the weeks of treatment (6 of 12 weeks). A weekly stool frequency response is defined as a stool frequency increase of 1 or more CSBMs per week compared with baseline, with abdominal pain unchanged or improved compared with baseline.
Time Frame: After completing 12-week course of SYN-010
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 20
Participants | 4 | 6 | 9

4. Secondary Outcome: Proportion of Overall Abdominal Pain Intensity Responders During the 12-week Treatment Period
Description: An overall abdominal pain intensity responder is defined as a patient with a weekly abdominal pain intensity response in at least 50% of the weeks of treatment (6 of 12 weeks). A weekly response abdominal pain intensity response is defined as a decrease in the patient's weekly average score for worst abdominal pain in the past 24 hours of at least 30% compared to baseline, with stool frequency unchanged or improved compared with baseline.
Time Frame: After completing 12-week course of SYN-010
Population: secondary outcomes measures were not analyzed as interim analysis showed that the study has not met its primary end point and the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 20
Participants | 4 | 4 | 7

5. Secondary Outcome: Proportion of Overall Bloating Responders During the 12-week Treatment Period
Description: An overall bloating responder is defined as a patient with a weekly bloating response in at least 50% of the weeks of treatment (6 of 12 weeks). A weekly bloating response is defined as a weekly average bloating score of at least 30% improvement compared to baseline, with stool frequency unchanged or improved compared with baseline.
Time Frame: After completing 12-week course of SYN-010
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 20
Participants | 3 | 3 | 1

6. Secondary Outcome: Proportion of Patients Using Rescue Medication
Description: Subjects will record their use of rescue medication throughout the study period. Proportion of patients using rescue medication after completing the 12-week course of treatment will be compared to those reporting usage at baseline screening period.
Time Frame: After completing 12-week course of SYN-010
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 20
Participants | 9 | 11 | 8

7. Other Pre Specified Outcome: Proportion of Patients With Adequate Relief
Description: Outcome will be assessed by evaluating proportion of patients reporting adequate relief pre- and post-treatment on validated questionnaire.
Time Frame: After completing 12-week course of SYN-010
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 17 | 14 | 18
Participants | 1 | 2 | 6

8. Other Pre Specified Outcome: Mean Change From Baseline in the Area-under-the-curve (AUC) of Breath Methane Production, Based on the 120-minute Lactulose Breath Test.
Description: Change in exhaled methane level as a potential predictor of constipation improvement will be evaluated by comparing lactulose breath tests pre- and post-treatment.
Time Frame: After completing 12-week course of SYN-010
Measure: Mean (Standard Deviation); unit: particles per million * min
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 20
particles per million * min | -18.678 (51.000) | -20.137 (78.738) | -39.199 (76.518)

9. Other Pre Specified Outcome: Change From Baseline in Breath Methane Production Based on a Single-point Breath Methane Test
Description: Change in exhaled methane level as a potential predictor of constipation improvement will be evaluated by comparing single-point breath tests pre- and post-treatment.
Time Frame: After completing course of SYN-010
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: particles per million
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 20
particles per million | -22.623 (26.7900) | -4.785 (26.3392) | -10.081 (36.0877)

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | SYN-010 21 mg | SYN-010 42 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 4/19 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYN-010 21 mg (N=20) | SYN-010 42 mg (N=19) | Placebo (N=20)
Hemiplegic Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYN-010 21 mg (N=20) | SYN-010 42 mg (N=19) | Placebo (N=20)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3)
Metallic Taste, Paresthesia, Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal Pain, Bloating, Flatulence, Nausea, Indigestion (Gastrointestinal disorders) | 4 (6) | 1 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03763175/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT03763175/SAP_001.pdf